CLINICAL TRIAL: NCT06283693
Title: The Effect of Mindfulness-based Stress Reduction Programme Given to Infertile Women on Perceived Stress, Anxiety, Depression and Cortisol Levels
Brief Title: The Effect of Mindfulness-based Stress Reduction Programme Given to Infertile Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, assoc. prof. dr, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RojdaBAYARYILDIRIM
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Depression Anxiety Disorder; Demography, Family; Awakening Early
Keywords: Infertility; women,; mindfulness; cortisol; anxiety; depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Infertility; Anxiety Disorders; Depression | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Randomized controlled classical experimental study
Who Masked: Participant
Masking Description: Computer-assisted randomization will be used in the study, and participants will be randomized to an intervention or control list control group in a 1:1 ratio by entering the number of samples to be reached through the program whose URL address is https://www.randomizer.org. Women who apply to the infertility outpatient clinic by the researcher and volunteer for the study who meet the sample selection criteria will be given numbers according to the order of outpatient clinic registration. A randomization sequence will be created according to these numbers and women will be assigned to the intervention and control groups by computer-assisted randomization. Since the study is a thesis, blinding will not be possible due to its nature.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimantal group: (Experimental): Intervention Group : The women in this group will receive a 4-week Mindfulness-Based Stress Reduction program in addition to routine outpatient clinic follow-up at the relevant institution. Before the implementation of the Mindfulness-Based Stress Reduction program, the women in the intervention group will be administered the Informed Voluntary Consent Form, Descriptive Characteristics Information Form, Perceived Stress Scale, DASS-21 and salivary cortisol measurements for pre-test measurements. After the mindfulness program, follow-up tests will be conducted in the 4th week. In the 8th week, the post-test will be conducted. In the post-test and follow-up test; Perceived Stress Scale, DASS-21 and salivary cortisol measurements will be applied.
  Interventions: Other: mindfulness-based stress reduction
- Control group: (No Intervention): The women in this group will not be subjected to any intervention and will be followed up in the routine outpatient clinic of the relevant institution. Informed Voluntary Consent Form, Descriptive Characteristics Information Form, Perceived Stress Scale, DASS-21 and salivary cortisol measurements will be applied for the pre-test measurements of the control group women. In the study, post-test measurements will be made 4 weeks after the pre-test measurements of the control group and follow-up measurements will be made 8 weeks later. Perceived Stress Scale, DASS-21 and salivary cortisol measurements will be applied to the women in the control group for pre-test, post-test and follow-up measurements.

INTERVENTIONS:
Other: mindfulness-based stress reduction — Müdahale grubundaki kadınlara depresyon, anksiyete ve stres düzeylerini azaltmak için farkındalık temelli bir stres azaltma programı uygulanacaktır. Program, haftada bir seans olmak üzere haftada iki kez toplam 4 hafta boyunca 8 seanstan oluşacaktır. Müdahale grubu haftada 2 seans alacaktır. Her seans 80 dakika sürecektir. Çalışmadaki seanslar, katılımcıların iş yoğunluğu, hayattaki sorumlulukları ve 4 hafta boyunca düzenli olarak katılamama ihtimalleri göz önünde bulundurularak zoom programı üzerinden gerçekleştirilecektir. 4 hafta/8 oturumluk MBSR programı tamamlandıktan sonra müdahale grubundaki kadınlara veri toplama formları tekrar uygulanacak ve son test ölçümleri yapılacaktır. Son test ölçümlerinden sonra müdahale grubundaki kadınların takip ölçümleri ölçümlerden 8 hafta sonra yapılacaktır.
  Arms: Experimantal group:

SUMMARY:
Purpose of the Study This study aims to determine the effect of mindfulness-based stress reduction program given to infertile women on perceived stress, anxiety, depression and salivary cortisol.

Materials and Method It will be conducted in a randomized controlled experimental design. This randomized controlled trial will follow the Consolidated Standards of Reporting Trials (CONSORT) 2010 guidelines.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled experimental study to determine the effect of mindfulness-based stress reduction program given to infertile women on perceived stress, anxiety, depression and salivary cortisol levels. It will be conducted in a randomized parallel controlled experimental design using Consolidated Standards of Reporting Trials (CONSORT) guidelines. Women applying to the infertility outpatient clinic of Health Sciences University Ümraniye Training and Research Hospital in Ümraniye district of Istanbul province will constitute the sample population of the study. Women applying to the infertility outpatient clinic who meet the inclusion criteria and who voluntarily agree to participate in the study will be included in the study. According to the power analysis, a total of 86 infertile women, 43 in the intervention group and 43 in the control group, will constitute the sample of the study. While Mindfulness-Based Stress Reduction Program will be applied to the intervention group with the zoom program, which is an online training platform, routine follow-up will be applied to the control group within the scope of outpatient follow-up of the relevant institution. The participants included in the study will be administered the Informed Voluntary Consent Form, Descriptive Characteristics Information Form, DASS-21, Perceived stress scale and Salivary cortisol test as part of the pre-test. Within the scope of post-test and follow-up test, DASS-21, Perceived stress scale and Salivary cortisol test will be applied again.

Discussion and conclusions of the study will be written as a result of the findings

ELIGIBILITY:
Inclusion Criteria:

* - Agree to participate in the 8-week MBSR training
* Having completed the Informed Consent Form and volunteering to participate in the study
* Speaking and understanding Turkish
* Idiopathic infertile women
* Primary infertile women
* YTU treatment has not started
* Having attempted YTU at most three times before
* Be able to use ZOOM program

Exclusion Criteria:

* - Illiteracy,
* The woman has a cognitive and auditory problem,
* Having a chronic disease
* Not having a psychiatric diagnosis (schizophrenia, bipolar disorder, major depression, anxiety disorders, etc.)
* Having participated in any awareness-based training program in the last 1 year

Exclusion Criteria

- Not participating in any session of the 8-session training program, not participating in any of the Pre-test, Post-test-1 and Post-test-2

Being an infertile woman

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Being an infertile woman
Enrollment: 84 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Informed Voluntary Consent Form (Annex 1) | Before implementation
  This form, which was created by the researchers, includes information about the intervention and control groups, explaining the content and purpose of the study to the participants, the time of the weekly program and how many days the program will last, when the research will end, which data collection tools will be used, for what purpose the data will be used, how information privacy will be ensured, the information of the researcher, and the consent of the participants and their voluntariness.
Identifying Characteristics Information Form (Annex 2) | Before implementation
  This form, prepared by the researchers in line with the literature, consists of 20 items. In addition to socio-demographic information such as age, education level, occupation, marriage duration, infertility history is questioned (Garland et al., Domar 2008; Sherratt & Lunn, 2013, Ozan & Okumuş, 2013, Güngör & Bejı̇ , 2015; Fanning et al., 2018;, ; Hosseini et al., 2020;; Örüklü, 2020).
Perceived Stress Scale (Appendix 3): | Before implementation
  The Perceived Stress Scale was developed as a five-point Likert-type rating scale with 14 items. The scale consists of "never (0), almost never" (1), "sometimes" (2), "often" (3) and "very often" (4) options. In this 14-item form, items 4-5-6-7-9-10 and 13 are reverse scored. The lowest and highest scores that a participant can obtain from this scale are 0 and 56, respectively. A high total score means a high Perceived Stress Level Scale. It can be said that participants with a score range between 0 and 35 have a positive stress level, can cope with stress effectively and the coping mechanisms they use are functional. It can be said that the methods used by the participants with a score range between 36-56 are not functional and therefore they cannot cope with stress effectively.
Depression-Anxiety-Stress Scale (Appendix 4) | Before implementation
  The Cronbach's alpha internal consistency coefficients of the 3 sub-dimensions of the scale were tested as .84 for the anxiety sub-dimension, .91 for the depression sub-dimension and .90 for the stress sub-dimension. The scale is a 4-point Likert-type form for self-assessment. The sub-dimensions and item distribution are as follows: Depression: 7 items in total, including items 3, 5, 10, 13, 16, 17 and 21. Anxiety: 2., 4., 7., 9., 15., 19. and 20. Stress: 1st, 6th, 8th, 11th, 12th, 14th and 18th items, totaling 7 items. In the internal consistency calculations of the scale, the Cronbach Alpha coefficient of the depression sub-dimension was .67; the Cronbach Alpha coefficient of the anxiety sub-dimension was .86; the Cronbach Alpha coefficient of the stress sub-dimension was .67 and the Cronbach Alpha coefficient for the whole scale was .87. There were no reverse items in the scale.
Collection and study of salivary cortisol samples | Before implementation
  For the determination of cortisol level; salivary cortisol measurement will be taken from the women in the intervention and control groups for the first test. Then, after the 4 -week MBSR program, salivary cortisol will be taken again from the intervention and control groups for the post-test. Then salivary cortisol test will be taken for follow-up at the 12th week. Saliva samples will be collected by the researcher. In our study, DRG brand Salivary tubes made of polypropylene (PP) / low density polyethylene (LD-PE) material especially designed for cortisol will be used for the collection and storage of saliva samples (Figure 1). These tubes provide high analytical performance from small volumes of samples. Patients will be asked to wet the cotton ball in the salivary tube (Figure 2) completely with saliva by holding it in their mouth for one minute. The samples will be refrigerated and centrifuged at 4000 g for 10 minutes in the biochemistry laboratory.

SECONDARY OUTCOMES:
Perceived Stress Scale (Appendix 3): | After the implemantation (4. week)
  The Perceived Stress Scale was developed as a five-point Likert-type rating scale with 14 items. The scale consists of "never (0), almost never" (1), "sometimes" (2), "often" (3) and "very often" (4) options. In this 14-item form, items 4-5-6-7-9-10 and 13 are reverse scored. The lowest and highest scores that a participant can obtain from this scale are 0 and 56, respectively. A high total score means a high Perceived Stress Level Scale. It can be said that participants with a score range between 0 and 35 have a positive stress level, can cope with stress effectively and the coping mechanisms they use are functional. It can be said that the methods used by the participants with a score range between 36-56 are not functional and therefore they cannot cope with stress effectively.
Depression-Anxiety-Stress Scale (Appendix 4) | After the implemantation (4. week)
  The Cronbach's alpha internal consistency coefficients of the 3 sub-dimensions of the scale were tested as .84 for the anxiety sub-dimension, .91 for the depression sub-dimension and .90 for the stress sub-dimension. The scale is a 4-point Likert-type form for self-assessment. The sub-dimensions and item distribution are as follows: Depression: 7 items in total, including items 3, 5, 10, 13, 16, 17 and 21. Anxiety: 2., 4., 7., 9., 15., 19. and 20. Stress: 1st, 6th, 8th, 11th, 12th, 14th and 18th items, totaling 7 items. In the internal consistency calculations of the scale, the Cronbach Alpha coefficient of the depression sub-dimension was .67; the Cronbach Alpha coefficient of the anxiety sub-dimension was .86; the Cronbach Alpha coefficient of the stress sub-dimension was .67 and the Cronbach Alpha coefficient for the whole scale was .87. There were no reverse items in the scale.
Collection and study of salivary cortisol samples | After the implemantation (4. week)
  For the determination of cortisol level; salivary cortisol measurement will be taken from the women in the intervention and control groups for the first test. Then, after the 4 -week MBSR program, salivary cortisol will be taken again from the intervention and control groups for the post-test. Then salivary cortisol test will be taken for follow-up at the 12th week. Saliva samples will be collected by the researcher. In our study, DRG brand Salivary tubes made of polypropylene (PP) / low density polyethylene (LD-PE) material especially designed for cortisol will be used for the collection and storage of saliva samples (Figure 1). These tubes provide high analytical performance from small volumes of samples. Patients will be asked to wet the cotton ball in the salivary tube (Figure 2) completely with saliva by holding it in their mouth for one minute. The samples will be refrigerated and centrifuged at 4000 g for 10 minutes in the biochemistry laboratory.

OTHER OUTCOMES:
Perceived Stress Scale (Appendix 3): | After the implemantation (8. week)
  The Perceived Stress Scale was developed as a five-point Likert-type rating scale with 14 items. The scale consists of "never (0), almost never" (1), "sometimes" (2), "often" (3) and "very often" (4) options. In this 14-item form, items 4-5-6-7-9-10 and 13 are reverse scored. The lowest and highest scores that a participant can obtain from this scale are 0 and 56, respectively. A high total score means a high Perceived Stress Level Scale. It can be said that participants with a score range between 0 and 35 have a positive stress level, can cope with stress effectively and the coping mechanisms they use are functional. It can be said that the methods used by the participants with a score range between 36-56 are not functional and therefore they cannot cope with stress effectively.
Depression-Anxiety-Stress Scale (Appendix 4) | After the implemantation (8. week)
  The Cronbach's alpha internal consistency coefficients of the 3 sub-dimensions of the scale were tested as .84 for the anxiety sub-dimension, .91 for the depression sub-dimension and .90 for the stress sub-dimension. The scale is a 4-point Likert-type form for self-assessment. The sub-dimensions and item distribution are as follows: Depression: 7 items in total, including items 3, 5, 10, 13, 16, 17 and 21. Anxiety: 2., 4., 7., 9., 15., 19. and 20. Stress: 1st, 6th, 8th, 11th, 12th, 14th and 18th items, totaling 7 items. In the internal consistency calculations of the scale, the Cronbach Alpha coefficient of the depression sub-dimension was .67; the Cronbach Alpha coefficient of the anxiety sub-dimension was .86; the Cronbach Alpha coefficient of the stress sub-dimension was .67 and the Cronbach Alpha coefficient for the whole scale was .87. There were no reverse items in the scale.
Collection and study of salivary cortisol samples | After the implemantation (8. week)
  For the determination of cortisol level; salivary cortisol measurement will be taken from the women in the intervention and control groups for the first test. Then, after the 4 -week MBSR program, salivary cortisol will be taken again from the intervention and control groups for the post-test. Then salivary cortisol test will be taken for follow-up at the 12th week. Saliva samples will be collected by the researcher. In our study, DRG brand Salivary tubes made of polypropylene (PP) / low density polyethylene (LD-PE) material especially designed for cortisol will be used for the collection and storage of saliva samples (Figure 1). These tubes provide high analytical performance from small volumes of samples. Patients will be asked to wet the cotton ball in the salivary tube (Figure 2) completely with saliva by holding it in their mouth for one minute. The samples will be refrigerated and centrifuged at 4000 g for 10 minutes in the biochemistry laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: YASEMİN AYDIN KARTAL, Doc. Dr., Principal Investigator — Health S.; ROJDA BAYAR YILDIRIM, PhD StD., Study Chair — Research H.; İBRAHİM KALE, Doc. Dr., Study Chair — Research H.
Locations (1):
- Saglık Bilimleri Universitesi, Istanbul, Turkey (Türkiye)